CLINICAL TRIAL: NCT01579630
Title: An Open Label, Randomized, Multicenter, Phase II Study to Compare Efficacy and Safety of Gefitinib/ Pemetrexed With Pemetrexed Alone as Maintenance Therapy in Patients With Advanced (Stage IV) EGFR Mutation Negative or T790M Single Mutation Nonsquamous NSCLC Who Respond to 4 Cycles of Pemetrexed/ Platinum as First-line Therapy
Brief Title: Genius Study Study to Compare Efficacy and Safety of Gefitinib/ Pemetrexed With Pemetrexed Alone as Maintenance Therapy in Patients With Stage IV EGFR Mutation Negative or T790M Single Mutation Who Respond to Pemetrexed/ Platinum as First-line Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taiwan University Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); Dalin Tzu Chi General Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator; Chief of Section of Thoracic Oncology of the Chest Department, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7913L00077
Record Dates: First submitted 2012-04-12; First posted 2012-04-18 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: NSCLC
Keywords: NSCLC; Nonsquamous; Maintenance therapy
MeSH Terms: interventions — Pemetrexed; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed 500mg/m2 iv (Experimental)
  Interventions: Drug: Pemetrexed 500mg/m2 iv
- Pemetrexed 500 mg/m2 i.v. and Gefitinib 250 mg (Experimental)
  Interventions: Drug: Pemetrexed 500mg/m2 iv and Gefitinib 250 mg

INTERVENTIONS:
Drug: Pemetrexed 500mg/m2 iv — EGFR mutation negative patients who continuously respond (CR, PR or SD) to the 4th cycle of pemetrexed/ cisplatin or pemetrexed/carboplatin will be randomized in a 1:1 ratio to receive either gefitinib/ pemetrexed, or pemetrexed alone as maintenance therapy until progression of disease (PD) or discontinuation of treatment for other reasons.
  Arms: Pemetrexed 500mg/m2 iv
Drug: Pemetrexed 500mg/m2 iv and Gefitinib 250 mg — EGFR mutation negative patients who continuously respond (CR, PR or SD) to the 4th cycle of pemetrexed/ cisplatin or pemetrexed/carboplatin will be randomized in a 1:1 ratio to receive either gefitinib/ pemetrexed, or pemetrexed alone as maintenance therapy until progression of disease (PD) or discontinuation of treatment for other reasons.
  Arms: Pemetrexed 500 mg/m2 i.v. and Gefitinib 250 mg

SUMMARY:
The study aims to randomize 52 patients with advanced (Stage IV) EGFR mutation negative nonsquamous non-small cell lung cancer (NSCLC) who respond (CR/PR/SD) to 4 cycles of pemetrexed / cisplatin or pemetrexed/carboplatin as first-line therapy. In order to achieve that, approximately 144 treatment naïve patients with advanced nonsquamous NSCLC need to be enrolled from around 6 investigational sites in Taiwan that have expertise in lung cancer diagnosis.

DETAILED DESCRIPTION:
The hypothesis tested in this study is that gefitinib / pemetrexed as maintenance therapy in patients with advanced (stage IV) EGFR mutation negative nonsquamous NSCLC who respond to 4 cycles of pemetrexed / cisplatin or pemetrexed/carboplatin as first-line therapy will achieve longer PFS than pemetrexed alone. We assume a median PFS of 4 months for patients receiving pemetrexed alone and the hazard ratio of pemetrexed alone compared to gefitinib/pemetrexed would be 0.42. It also indicates that the median PFS in gefitinib/pemetrexed group will be approximately 9.52 months. This is a 2-arm study in a 1:1 randomisation. Assuming an uniform accrual of 12-month with an addition of 12-month follow-up period, the total evaluable number of patients will be 52 to achieve a power of 80% and one-sided significance level of 0.025 to detect such difference between gefitinib/pemetrexed and pemetrexed alone.

Assuming 60% of patients respond (CR/PR/SD) to 4 cycles of pemetrexed/gefitinib, and among them 60% are EGFR mutation negative, 144 patients need to be enrolled to receive 4 cycles of pemetrexed/cisplatin or pemetrexed/carboplatin as first-line therapy.

Besides, the result of anaplastic lymphoma kinase gene (ALK) mutation will be retrospectively collected if the mutation is available for study patients during the study period.

ELIGIBILITY:
Inclusion Criteria summary

1. Provision of written informed consent
2. Patients age 20 years or older
3. Histological or cytological confirmed advanced (stageIV) nonsquamous NSCLC
4. NSCLC treatment naïve(except patients who have pre- and post-operative non-platinum based adjuvant chemotherapy greater than 6 months prior to enrolment can be enrolled.)
5. Measurable disease according to RECIST (Version 1.1) criteria
6. World Health Organization (WHO) performance status (PS) of 0 to 1
7. Provision of cancer tissue sample for mutation testing or the result of EGFR mutation test is negative (single T790M mutation positive patients can also be enrolled)

Exclusion Criteria summary

1. Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
2. Known severe hypersensitivity to gefitinib, pemetrexed, cisplatin and carboplatin or any of the excipients of these products
3. Known severe hypersensitivity to pre-medications required for treatment with pemetrexed / cisplatin or pemetrexed/carboplatin doublet chemotherapy
4. Absolute neutrophil counts (ANC) less than 2.0 x 109/L (2,000/mm3), platelets less than 100 x 109/L (100,000/mm3) or haemoglobin less than 10 g/dl
5. Pre-existing idiopathic pulmonary fibrosis evidence by CT scan at baseline
6. Serum bilirubin is greater than 1.5 times the upper limit of reference range
7. Serum creatinine is greater than 1.5 times the ULRR
8. Unable to tolerate pemetrexed/ cisplatin or pemetrexed/carboplatin doublet chemotherapy, as judged by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 4 months
  Progression of disease will be calculated from the tumour measurements collected at each tumour assessment per the RECIST (V1.1) criteria and/or the date of patient death.

SECONDARY OUTCOMES:
Overall objective tumour response | up to 1 year
  The RECIST (V1.1) criteria will be used to assess objective tumour response. Details of target and non-target lesions will be collected on the appropriate CRF pages and used to calculate tumour response. Post-baseline tumour evaluations should use the same modality (CT scan or magnetic resonance imaging [MRI]) as used at baseline and should preferably be undertaken at the same institution.

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans General Hospital -Taipei, Taipei, Taiwan